CLINICAL TRIAL: NCT04926610
Title: The Effect of Proactive Clinical Ethics Consultations on End-of-life Care of the Critically Ill in the Intensive Care Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUH-IRB-20130379
Record Dates: First submitted 2021-02-21; First posted 2021-06-15 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Proactive Clinical Ethics Consultation; the Critically Ill
Keywords: proactive clinical ethics consultation; critically ill; end-of-life care; interprofessional practicethe; interprofessional education
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proactive clinical ethics consultation group (Experimental)
  Interventions: Other: proactive clinical ethics consultation
- routine care group (No Intervention)

INTERVENTIONS:
Other: proactive clinical ethics consultation — When the patients meet the initiation criteria of this study, the patients were randomly assigned to the intervention group (providing proactive clinical ethics consultation) and the routine care group (no proactive clinical ethics consultation) after obtaining the consent of the subjects.
  Arms: proactive clinical ethics consultation group

SUMMARY:
Study objective: This study is planning to explore factors predicting the use of life-sustaining treatment, develop the screening criteria of proactive clinical ethics consultations, the effect of proactive clinical ethics consultations and interprofessional practice on end-of-life care of the critically ill in the intensive care settings, and develop the competency for trainees by interprofessional education.

Methods: Data will be collected prospectively. Data between January 2013 and April 2014 was collected from hospital electronic record and ethics consultation document. All data will be analyzed for patients dying in the intensive care settings during the first stage of the study. Factors predicting the use of life-sustaining treatment will be determined. The Delphi technique will be applied to secure a consensus among the panel of experts chosen to help develop the screening criteria of proactive ethics consultations. A prospective randomized controlled trial will be conducted during the second stage of the study on a convenience sample of adult critical ill patients in the intensive care settings. Patients will randomize to the intervention group receive proactive ethics consultations. The control group will undergo routine intensive care, receiving clinical ethics consultations as requested by healthcare team, patients or family. All participants will be asked to complete a questionnaire rating their satisfaction with the healthcare process and consultations if conducted. Mean length of stay and the duration of the use of life-sustaining treatment will be compared between two groups. Secondary outcomes will include the proportion of satisfied families and healthcare team members. The interprofessional education with the core curriculum and case scenario for simulation will be developed, implement, and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Medical staff involved in caring for terminal patients
2. Cases of active clinical ethics consultation in our hospital

Exclusion Criteria:

1. Medical staff who refuse to participate in the study or are unable to understand the way the study is conducted
2. Cases of refusing to participate in the research or unable to understand the way the research is conducted.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2014-04-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
hospital length of stay | through study completion, an average of 2 years
  days that patient in the hospital
ICU length of stay | through study completion, an average of 2 years
  days that patient in the intensive care unit
use of life-sustaining treatment | through study completion, an average of 2 years
  days of the use of life-sustaining treatment

SECONDARY OUTCOMES:
family or surrogate satisfaction questionnaire | within 4 weeks after patient discharge
  family or surrogate satisfaction for ethics consultation
family or surrogate satisfaction questionnaire | within 4 weeks after patient discharge
  family or surrogate satisfaction for patient care
healthcare provider satisfaction questionnaire | within 2 weeks after patient discharge
  healthcare provider satisfaction for ethics consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Lin YK, Chen CW, Yeh YS, Lin CJ, Huang YW, Lin YC, Sheu CC. Impacts of mandatory clinical ethics consultation on resource utilization and ethical conflicts in critically ill patients: a comparison between medical and surgical intensive care units. BMC Med Ethics. 2025 Aug 2;26(1):110. doi: 10.1186/s12910-025-01268-4. PMID 40753248